CLINICAL TRIAL: NCT03421327
Title: Genetic Risk: Whether, When, and How to Tell Adolescents
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00121662; R01HG008045 (NIH)
Record Dates: First submitted 2018-01-02; First posted 2018-02-05 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Huntington Disease; Hereditary Breast and Ovarian Cancer; Hereditary Cancer; Hereditary Non-polyposis Colon Cancer; Hereditary Non-Polyposis Colorectal Cancer Syndrome
MeSH Terms: conditions — Huntington Disease; Hereditary Breast and Ovarian Cancer Syndrome; Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Families at-risk for HD: No interventions will be administered. Participation involves one semi-structured interview that will last up to one hour. The interview will be scheduled at a time and place that is convenient for the participant. The participant will be given the option to conduct the interview via phone, Skype, or in-person at Johns Hopkins.
- Families at-risk for hereditary cancer: No interventions will be administered. Participation involves one semi-structured interview that will last up to one hour. The interview will be scheduled at a time and place that is convenient for the participant. The participant will be given the option to conduct the interview via phone, Skype, or in-person at Johns Hopkins.
- Genetic Counselors: No interventions will be administered. Participation involves one semi-structured interview that will last up to one hour. The interview will be scheduled at a time and place that is convenient for the participant. The participant will be given the option to conduct the interview via phone, Skype, or in-person at Johns Hopkins.

SUMMARY:
This study is being conducted to learn more about family communication of genetic risk information. Semi-structured interviews lasting up to one hour will be conducted with three populations: parent/child pairs at risk for Huntington's Disease, parent/child pairs at risk for hereditary cancer, and genetic counselors.

DETAILED DESCRIPTION:
The investigators currently lack an adequate understanding of how parents and children feel about genetic risk/status, how it is communicated, and how it influences wellbeing and family relationships. This understanding is vital in order for genetic counselors and other health care professionals to provide the best guidance possible to families. However, little research has been conducted on the impact of genetic risk information or testing on children from the perspective of the child. The research proposed here is uniquely positioned to help fill this gap.

For this study, the investigators will interview 15-20 parent/child pairs who are at risk for Huntington's Disease (HD), 15-20 parent/child pairs who are at risk for hereditary cancer, and 15-20 certified genetic counselors. Interviews will last no more than one hour and will be conducted at a time and place that is convenient for the participant. The investigators will offer participants a choice of conducting the interview in a private conference room at the Berman Institute of Bioethics, or remotely by Skype or telephone. Parents and children will be interviewed separately. Parents will be asked about the decision process behind how and when they disclosed genetic information to their child, style of family communication, advice for other parents in similar situations, and other questions related to the subject of communication of genetic information to minors. Children will be asked about their experience learning genetic risk information, style of family communication, how they felt, advice for other kids in similar situations, and other questions related to the subject of communication of genetic information to minors.

ELIGIBILITY:
Inclusion Criteria:

* Parents at-risk for HD, affected by HD, or be the spouse/partner of someone living who at risk for or affected by HD.
* Parents who have or have had a diagnosis of hereditary cancer, or the spouse/partner of someone living who has or has had had a diagnosis of hereditary cancer.
* Children ages 15-17 who are at risk for either HD or hereditary cancer

Exclusion Criteria:

* Parents and children who have not yet communicated about genetic risk
* Children younger than age 15

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include individuals who reside in the USA, speak English, and are able to participate in one interview either in person, via phone, or via Skype.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Qualitative analysis of how parents and children with either Huntington's Disease or hereditary cancer communicate about genetic risk information | 1.5 years
  Qualitative interview performed at one occasion where the patient describes when and how genetic risk information was disclosed to minor as well as perspectives from both parent and child.

CONTACTS AND LOCATIONS:
Overall Officials: Debra Mathews, PhD, MA, Principal Investigator — Johns Hopkins Berman Institute of Bioeithics
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith LA, Ullmann JF, Olson HE, Achkar CM, Truglio G, Kelly M, Rosen-Sheidley B, Poduri A. A Model Program for Translational Medicine in Epilepsy Genetics. J Child Neurol. 2017 Mar;32(4):429-436. doi: 10.1177/0883073816685654. Epub 2017 Jan 6. PMID 28056630
- [Background] Jarvik GP, Amendola LM, Berg JS, Brothers K, Clayton EW, Chung W, Evans BJ, Evans JP, Fullerton SM, Gallego CJ, Garrison NA, Gray SW, Holm IA, Kullo IJ, Lehmann LS, McCarty C, Prows CA, Rehm HL, Sharp RR, Salama J, Sanderson S, Van Driest SL, Williams MS, Wolf SM, Wolf WA; eMERGE Act-ROR Committee and CERC Committee; CSER Act-ROR Working Group; Burke W. Return of genomic results to research participants: the floor, the ceiling, and the choices in between. Am J Hum Genet. 2014 Jun 5;94(6):818-26. doi: 10.1016/j.ajhg.2014.04.009. Epub 2014 May 8. PMID 24814192
- [Background] Appelbaum PS, Parens E, Waldman CR, Klitzman R, Fyer A, Martinez J, Price WN 2nd, Chung WK. Models of consent to return of incidental findings in genomic research. Hastings Cent Rep. 2014 Jul-Aug;44(4):22-32. doi: 10.1002/hast.328. Epub 2014 Jun 11. PMID 24919982
- [Background] Garber JE, Offit K. Hereditary cancer predisposition syndromes. J Clin Oncol. 2005 Jan 10;23(2):276-92. doi: 10.1200/JCO.2005.10.042. PMID 15637391
- [Background] Quarrell OW, Rigby AS, Barron L, Crow Y, Dalton A, Dennis N, Fryer AE, Heydon F, Kinning E, Lashwood A, Losekoot M, Margerison L, McDonnell S, Morrison PJ, Norman A, Peterson M, Raymond FL, Simpson S, Thompson E, Warner J. Reduced penetrance alleles for Huntington's disease: a multi-centre direct observational study. J Med Genet. 2007 Mar;44(3):e68. doi: 10.1136/jmg.2006.045120. PMID 17361007
- [Background] Ford D, Easton DF, Stratton M, Narod S, Goldgar D, Devilee P, Bishop DT, Weber B, Lenoir G, Chang-Claude J, Sobol H, Teare MD, Struewing J, Arason A, Scherneck S, Peto J, Rebbeck TR, Tonin P, Neuhausen S, Barkardottir R, Eyfjord J, Lynch H, Ponder BA, Gayther SA, Zelada-Hedman M, et al. Genetic heterogeneity and penetrance analysis of the BRCA1 and BRCA2 genes in breast cancer families. The Breast Cancer Linkage Consortium. Am J Hum Genet. 1998 Mar;62(3):676-89. doi: 10.1086/301749. PMID 9497246
- [Background] McConkie-Rosell A, Spiridigliozzi GA, Melvin E, Dawson DV, Lachiewicz AM. Living with genetic risk: effect on adolescent self-concept. Am J Med Genet C Semin Med Genet. 2008 Feb 15;148C(1):56-69. doi: 10.1002/ajmg.c.30161. PMID 18200514
- [Background] Hamilton RJ. Using skype to conduct interviews for psychosocial research. Comput Inform Nurs. 2014 Aug;32(8):353-8. doi: 10.1097/CIN.0000000000000095. No abstract available. PMID 25133565
- [Background] Janghorban R, Latifnejad Roudsari R, Taghipour A. Skype interviewing: the new generation of online synchronous interview in qualitative research. Int J Qual Stud Health Well-being. 2014 Apr 15;9:24152. doi: 10.3402/qhw.v9.24152. eCollection 2014. PMID 24746247
- [Background] Meropol NJ, Daly MB, Vig HS, Manion FJ, Manne SL, Mazar C, Murphy C, Solarino N, Zubarev V. Delivery of Internet-based cancer genetic counselling services to patients' homes: a feasibility study. J Telemed Telecare. 2011;17(1):36-40. doi: 10.1258/jtt.2010.100116. Epub 2010 Nov 19. PMID 21097566
- [Background] Hilgart JS, Hayward JA, Coles B, Iredale R. Telegenetics: a systematic review of telemedicine in genetics services. Genet Med. 2012 Sep;14(9):765-76. doi: 10.1038/gim.2012.40. Epub 2012 Apr 12. PMID 22498847
- [Background] Abdolahi A, Bull MT, Darwin KC, Venkataraman V, Grana MJ, Dorsey ER, Biglan KM. A feasibility study of conducting the Montreal Cognitive Assessment remotely in individuals with movement disorders. Health Informatics J. 2016 Jun;22(2):304-11. doi: 10.1177/1460458214556373. Epub 2014 Nov 11. PMID 25391849
- [Background] Trondsen MV, Bolle SR, Stensland GO, Tjora A. Video-confidence: a qualitative exploration of videoconferencing for psychiatric emergencies. BMC Health Serv Res. 2014 Oct 31;14:544. doi: 10.1186/s12913-014-0544-y. PMID 25359404